CLINICAL TRIAL: NCT04095884
Title: An Observational Trial Designed to Elucidate the Pathways by Which Inflammation Contributes to Anaemia in Sick Rural African Children From 6 Months to 36 Months
Brief Title: An Observational Study Designed to Elucidate the Pathways by Which Inflammation Contributes to Anaemia in Sick Rural African Children From 6 Months to 36 Months
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: SCC 17097
Record Dates: First submitted 2019-09-04; First posted 2019-09-19 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Iron Deficiency, Anaemia in Children
MeSH Terms: conditions — Iron Deficiencies | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — samples will collected at baseline, day3 , day 7 and day 14
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Urinary Tract Infection: Inclusion criteria (one from the list below):
  1. Positive leukocytes, positive nitrites on dipstick
  2. Negative leukocytes, Positive nitrites on dipstick
  3. Positive leukocytes, negative nitrites, plus bacteriuria on microscopy
  4. Positive leukocytes, negative nitrities plus no bacteriuria, only pyuria on microscopy PLUS clinical features e.g. fever, pain on urination, offensive smelling urine.
  Exclusion criteria (one from the list below):
  1. No evidence of UTI on dipstick
  Interventions: Procedure: blood sampling
- Upper respiratory tract infection: Inclusion criteria (one from the list below)::
  1. Evidence of nasal discharge AND/OR
  2. Inflammation throat/ tonsils on direct examination AND/OR
  3. Inflammation of middle or outer ear on direct examination
  4. History of fever AND history of stridor/ barking cough
  5. History of fever AND lymphadenopathy AND/ OR URTI symptoms i.e sore throat/ cough
  Exclusion criteria (one from the list below)::
  1. Foreign body inserted in either nose/ ear
  2. Traumatic perforation of ear drum
  3. Allergic rhinitis i.e. good contact history
  4. Evidence of LRTI
  Interventions: Procedure: blood sampling
- Lower respiratory tract infection: Inclusion criteria (one from the list below):
  1. Focal signs on auscultation of the chest i.e crepitations/ wheeze/ reduced air entry
  2. Fever > 38.5C AND chest recessions AND/OR raised respiratory rate
  3. Radiological evidence of LRTI
  Exclusion criteria (one from the list below):
  1. Positive malaria test OR suspicion of metabolic acidosis causing tachypnoea and fever
  Interventions: Procedure: blood sampling
- Diarrhoea/ gastroenteritis: Inclusion criteria (one from the list below):
  1. Abrupt onset of 3 or more loose/liquid stools/ day
  2. Ova, cysts, parasites identified on stool microscopy PLUS symptomatic diarrhoea,and/ or fever and/or vomiting
  3. Fever AND vomiting WITHOUT other source of fever i.e UTI/LRTI/URTI
  Exclusion criteria (one from the list below):
  1. Normal breast milk stool
  2. Neurological cause of vomiting
  Interventions: Procedure: blood sampling

INTERVENTIONS:
Procedure: blood sampling — observational study and no intervention will be given. only blood samples collected and treated with iron supplements

SUMMARY:
The Investigator have previously shown that hepcidin is up-regulated even by low levels of inflammation and, according to our prior stable isotope studies, is predicted to block iron absorption. In this follow-up observational study, the investigator aim to characterise the relationship between infections, acute inflammation, hepcidin and iron iron deficiency anaemia in rural African children. The Investigator will study 200 sick children (6-36 months of age) living in the rural region of West Kiang.

The Investigator will:

1. Recruit 50 sick febrile children in each of 4 categories; Upper Respiratory tract infections, Lower respiratory tract infections (pneumonia), Urinary tract infections, gastroenteritis.
2. Assess iron absorption and its relationship to iron and anaemia status, inflammation, EPO, erythroferrone and hepcidin.

DETAILED DESCRIPTION:
Aim 1: To test whether non-malarial infections increase hepcidin levels and for how long in sick children (note that the investigator exclude malaria because the investigator and others have previously examined the effect of malaria).

Hypothesis 1: On day 0, 3 and 7 of acute illness, hepcidin will be higher when compared to levels in well children. On Day 14 iron absorption and hepcidin levels will have returned to baseline.

Research Question 1: What affect do non-malarial infections (upper respiratory tract infections, lower respiratory tract infections, urinary tract infections and gastroenteritis) have on hepcidin levels and how long does this effect last?

Aim 2: To retest our existing hepcidin threshold for discriminating iron absorbers from non-absorbers by repeating our prior ROC analysis based on a much larger sample.

Hypothesis: On day 0, 3 and 7 of acute illness, iron absorption will be lower. On Day 14, iron absorption will be equivalent to iron absorption in well children. Note that the Hepcidin levels and iron absorption data obtained in this study will be compared with the results obtained from similarly aged children in IDeA Study 1 (SCC 1664). Also note that The investigator anticipate that most of the children enrolled in this study will have a base-line level of anaemia (eg Hgb<11g/dL).

Research Question: What is the relationship between hepcidin and oral iron absorption in acute illness and convalescence and how does this differ from the relationship in well children?

Aim 3: To examine EPO synthesis and EPO resistance in children with acute non-malarial infections?

Hypotheses:

1. Children with acute non-malaria infections will have both acute and chronic anaemia of inflammation.
2. EPO is increased during acute infection.

Research Question: Is there decreased EPO synthesis and/or increased EPO resistance in children with acute non-malarial infections living in rural Gambia?

Aim 4: To examine erythroferrone in children with acute non-malarial infections leaving in rural Gambia.

Hypothesis: First The investigator will conduct a hypothesis-free exploratory analysis to assess whether erythroferrone behaves as predicted based upon mouse models (ie up-regulated by stress erythropoiesis and inversely related to hepcidin). The investigator additionally hypothesize that there may be a vicious cycle initiated by inflammation and then perpetuated by the consequent low levels of (iron-restricted) erythropoiesis, leading to low erythroferrone and loss of hepcidin suppression.

Research Question: What is the relationship between erythroferrone, iron status, inflammation, hepcidin, EPO and CRP in anaemic and non-anaemic children living in rural Gambia? This is an observational study of 200 sick children who will be recruited at the Keneba clinic. Each child will be seen four times (at day 0, 3, 7 14).

200 subjects aged 6 -36m brought to Keneba clinic with an acute illness. 50 patients from each category: Upper respiratory tract infections (including ear, nose and throat infections), Lower respiratory tract infections, urinary tract infections and gastroenteritis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female children ages 6-36 months
* Fever ( > 37.5C) and/or signs of illness.
* Signed or fingerprinted or personally marked written informed consent obtained from their parent/guardian.
* Parent/guardian plans for subject to reside in study site area and are able and willing to adhere to all protocol visits and procedures.

Exclusion Criteria:

1. Critically unwell requiring stabilisation and transfer i.e. scores 3 on initial assessment
2. Sickle cell disease
3. Evidence of hookworm infection by stool microscopy
4. Administration of immunosuppressants or other immune-modifying agents within 90 days prior to study IP administration (e.g., systemic corticosteroids at doses equivalent to ≥ 0.5 mg/kg/day of prednisone for more than 14 days; topical steroids including inhaled and intranasal steroids are not exclusionary).
5. Administration of systemic antibiotic treatment within 3 days prior to study enrolment.
6. Any history of or evidence for chronic clinically significant (as per investigator assessment) disorder or disease (including, but not limited to, immunodeficiency, autoimmunity, malnutrition*, congenital abnormality, bleeding disorder, and pulmonary, cardiovascular, metabolic, neurologic, renal, or hepatic disease). * Other than the exclusionary clinical diagnosis of malnutrition for all subjects, in children 2 to 5 years of age, malnutrition is also defined as a weight-for-height Z-score of less than -3 as per WHO reference standards.
7. Any history of human immunodeficiency virus, chronic hepatitis B or chronic hepatitis C infections.
8. Any condition that in the opinion of the investigator might compromise the safety or well-being of the subject or compromise adherence to protocol procedures
9. Participation in another MRC study

Ages: 6 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: sick children with fever
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-07-17 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Change in Serum hepcidin from baseline to day 14 | Day 14
Change in Clinical score of site and severity of infection and inflammation from baseline to day 14 | Day 14

SECONDARY OUTCOMES:
serum iron levels | Day 0, 3, 7 & 14
  Increase in serum iron levels above baseline following an oral ferrous fumarate dose as a measure of iron absorption
Erythropoietin | Day 0, 3, 7 & 14
Erythroferrone | Day 0, 3, 7 & 14

CONTACTS AND LOCATIONS:
Locations (1):
- Keneba MRC Unit, West Kiang, City of Banjul, The Gambia